CLINICAL TRIAL: NCT03080545
Title: An Open-Label, Study Evaluating Enstilar® (Calcipotriene and Betamethasone Dipropionate) Foam, 0.005%/0.064% QD in Psoriasis Patients Being Treated With Biologic Agents
Brief Title: Enstilar in Combination With Biologic Agents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC01
Record Dates: First submitted 2017-03-02; First posted 2017-03-15 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label Enstilar (Experimental): open label
  Interventions: Drug: Enstilar 0.005%-0.064% Topical Foam

INTERVENTIONS:
Drug: Enstilar 0.005%-0.064% Topical Foam — Topical foam

SUMMARY:
Patients receiving biologic therapy with 5% or less body surface area will receive Enstilar topical foam for 16 weeks.

DETAILED DESCRIPTION:
A two-phase, single center, observational study of 25 subjects to assess 4 weeks of adjunctive therapy of Enstilar® QD followed by 12 weeks QD on two consecutive days a week to patients with ≤5% BSA who are receiving biologic therapy for at least 24 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults ≥ 18 years of age.
2. Diagnosis of chronic plaque-type psoriasis.
3. Able to give written informed consent prior to performance of any study related procedures.
4. Treated with a biologic agent for a minimum of 24 weeks at baseline.
5. Plaque-type psoriasis as defined at screening and baseline by BSA ≤ 5%.
6. Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options: hormonal contraception; intrauterine device (IUD); tubal ligation; or partner's vasectomy; Male or female condom diaphragm with spermicide, cervical cap with spermicide, or contraceptive sponge with spermicide.
7. Subject must be in general good health (except for psoriasis) as judged by the Investigator, based on medical history, physical examination.

Exclusion Criteria:

1. >5% Body Surface Area
2. Any condition, which would place the subject at unacceptable risk if he/she were to participate in the study.
3. Pregnant or breast feeding, or considering becoming pregnant during the study.
4. Use of any investigational drug within 4 weeks prior to randomization, or within 5 pharmacokinetic/pharmacodynamic half lives, if known (whichever is longer).
5. Use of oral systemic medications for the treatment of psoriasis within 4 weeks (includes, but not limited to, oral corticosteroids, methotrexate, acitretin, apremilast and cyclosporine).
6. Patient used other topical therapies to treat within 2 weeks of the Baseline Visit (includes, but not limited to, topical corticosteroids, vitamin D analogs, or retinoids).
7. Patient received UVB phototherapy within 2 weeks of Baseline.
8. Patient received PUVA phototherapy within 4 weeks of Baseline.
9. Patient has a known hypersensitivity to the excipients of Enstilar® as stated in the label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Physician global assessment multiplied by body surface area improvement after 16 weeks of Enstilar® adjunctive therapy | 16 weeks
  pga x bsa

SECONDARY OUTCOMES:
Physician Global Assessment | 16 weeks
  PGA
Body Surface area | 16 weeks
  BSA
dermatology life quality index; TSQ-9 Treatment Satisfaction Questionnaire | 16 weeks
  satisfaction determined by patient reported outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No